CLINICAL TRIAL: NCT02281032
Title: Informed Palliative Care in Nursing Homes Through the interRAI Palliative Care Instrument: A Study Protocol Based on the Medical Research Council Framework
Brief Title: Informed Palliative Care in Nursing Homes Through the interRAI Palliative Care Instrument
Acronym: interRAI PC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: KU Leuven (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); University Ghent (Other); Vrije Universiteit Brussel (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Kirsten Hermans, KU Leuven, LUCAS, KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBO-IWT 100036; S56798 (Registry Identifier: Medical Ethics Committee UZ KU Leuven)
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Nursing Home Residents With Palliative Care Needs
Keywords: Palliative Care; Nursing Homes; interRAI Palliative Care instrument; Older adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interRAI Palliative Care (Other): 15 experimental nursing homes:
  * Caregivers of 15 participating nursing homes receive a training about the interRAI PC and the BelRAI webapplication
  * Caregivers of 15 experimental nursing homes fill out the interRAI PC multidisciplinary every three months during one year for all nursing home residents with palliative care needs. Based on the results (Client Assessment Protocols and Scales) of the interRAI PC instrument, care plans are being evaluated, adapted and designed.
  Interventions: Other: interRAI PC
- No interRAI Palliative Care (No Intervention): 15 control nursing homes:
  - Caregivers of control nursing homes do not receive the intervention and provide care as usual

INTERVENTIONS:
Other: interRAI PC — PREPARATORY PHASE
  * Step 0: Introductory information
  * Step 1: Training on the interRAI PC and the BelRAI webapplication
  * Step 2: Introduction on the interRAI PC and the BelRAI webapplication in the organization
  IMPLEMENTATION PHASE
  * Step 3: Identification of residents with palliative care needs, based on the surprise question
  * Step 4: Informed consent signature requirements
  * Step 5: Login to the BelRAI webapplication
  * Step 6: Definitions of roles and functions
  * Step 7: Completion of the interRAI PC
  * Step 8: Interpretation of results
  * Step 9: Use of results
  Other Names: FLIECE-interRAI PC
  Arms: interRAI Palliative Care

SUMMARY:
BACKGROUND Nursing homes are important locations for palliative care. Through comprehensive geriatric assessments (CGAs), evaluations can be made of the palliative care needs of nursing home residents. The interRAI Palliative Care instrument (interRAI PC) is a CGA that evaluates diverse palliative care needs of adults in all healthcare settings. The evaluation results in Client Assessment Protocols (CAPs: indications of problems that need addressing) and Scales (e.g. Palliative Index for Mortality (PIM)) which can be used to design, evaluate and adjust care plans. This study aims to examine the effect of using the interRAI PC on the quality of palliative care in nursing homes. Additionally, it aims to evaluate the feasibility and validity of the interRAI PC.

METHODS This study covers phases 0, I and II of the Medical Research Council (MRC) framework for designing and evaluating complex interventions, with a longitudinal, quasi-experimental pretest-posttest design and with mixed methods of evaluation. In phase 0, a systematic literature search is conducted. In phase I, the interRAI PC instrument is adapted for use in Belgium and implemented on the BelRAI-website and a practical training is developed. In phase II, the intervention is tested in fifteen nursing homes. Participating nursing homes fill out the interRAI PC during one year for all residents receiving palliative care. Using a pretest-posttest design with quasi-random assignment to the intervention or control group, the effect of the interRAI PC on the quality of palliative care is evaluated with the Palliative care Outcome Scale (POS). Psychometric analysis is conducted to evaluate the predictive validity of the PIM and the convergent validity of the CAP 'Mood' of the interRAI PC. Qualitative data regarding the usability and face validity of the instrument are collected.

DISCUSSION This is the first study to evaluate the validity and effect of the interRAI PC in nursing homes, following a methodology based on the MRC framework. This approach improves the study design and implementation and will contribute to a higher generalizability of results. The final result will be a psychometrically evaluated CGA for nursing home residents receiving palliative care.

ELIGIBILITY:
Inclusion Criteria:

* 65+
* residing in a nursing home
* having palliative care needs (based on the 'surprise question': 'would you be surprised if this person was to die within 6 to 12 months?') (Hubard G, 2011)

Exclusion Criteria:

* 65-
* not residing in a nursing home
* no palliative care needs

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
The effect of using the interRAI PC instrument on the quality of palliative care in nursing homes evaluated by the Palliative care Outcome Scale (POS) | 1 year
  Using a pretest-posttest design with quasi-random assignment to the intervention or control group, the effect of the interRAI PC on the quality of palliative care is evaluated with the Palliative care Outcome Scale (POS)

SECONDARY OUTCOMES:
The validity of the interRAI PC for use in nursing homes assessed by Psychometric analysis | 1 year
  Psychometric analysis is conducted to evaluate the predictive validity of the Palliative Index for Mortality (PIM) of the interRAI PC and the convergent validity of the CAP 'Mood' of the interRAI PC. Qualitative data regarding the face validity of the instrument are collected through focus groups, interviews and field notes
The feasibility of the interRAI C for use in nursing homes assessed through focus groups, interviews and field notes | 1 year
  Qualitative data regarding the feasibility of the instrument are collected through focus groups, interviews and field notes

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Hermans, Principal Investigator — KU Leuven, LUCAS; Nele Spruytte, Principal Investigator — KU Leuven, LUCAS; Joachim Cohen, Principal Investigator — End-of-Life Care Research Group, Vrije Universiteit Brussel (VUB) & Ghent University; Chantal Van Audenhove, Principal Investigator — KU Leuven, LUCAS; Anja Declercq, Principal Investigator — KU Leuven, LUCAS
Locations (1):
- KU Leuven, LUCAS, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Hermans K, De Almeida Mello J, Spruytte N, Cohen J, Van Audenhove C, Declercq A. A comparative analysis of comprehensive geriatric assessments for nursing home residents receiving palliative care: a systematic review. J Am Med Dir Assoc. 2014 Jul;15(7):467-476. doi: 10.1016/j.jamda.2014.01.002. Epub 2014 Feb 22. PMID 24569081
- [Derived] Hermans K, Spruytte N, Cohen J, Van Audenhove C, Declercq A. Informed palliative care in nursing homes through the interRAI Palliative Care instrument: a study protocol based on the Medical Research Council framework. BMC Geriatr. 2014 Dec 5;14:132. doi: 10.1186/1471-2318-14-132. PMID 25479633